CLINICAL TRIAL: NCT00133185
Title: A Randomized, Double-Blind, Parallel-Group Assessment of the Safety and Efficacy of Telmisartan 40mg Plus Hydrochlorothiazide 12.5 mg in Comparison With Losartan 50 mg Plus Hydrochlorothiazide 12.5 mg in Taiwanese Patients With Mild to Moderate Hypertension
Brief Title: A Randomized, Double-blind, Parallel-group Assessment of the Safety and Efficacy of Telmisartan 40mg Plus Hydrochlorothiazide 12.5mg (Micardis Plus) in Comparison With Losartan 50mg Plus Hydrochlorothiazide 12.5mg in Taiwanese Patients With Mild to Moderate Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.406
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide; Losartan

INTERVENTIONS:
Drug: telmisartan 40 mg/hydrochlorothiazide 12.5 mg
Drug: losartan 50 mg/hydrochlorothiazide 12.5 mg

SUMMARY:
The primary objective of this trial is to compare the efficacy and safety of telmisartan 40 mg/hydrochlorothiazide 12.5mg (Micardis Plus) with that of losartan 50 mg/hydrochlorothiazide 12.5 mg, a reference AIIA combined with diuretic, in Taiwanese patients with mild to moderate hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Mild to moderate hypertension as defined by a morning mean(>95 and <115mmHg) of two diastolic blood pressure measurements (DBP) after 5 min in the sitting position following a minimum 2-week placebo run in phase.Mean sitting systolic blood pressure (SBP) must be >140 and <200mmHg. The mean DBP and SBP values are calculated as the mean of the two sitting measurements taken 2 min apart just before the drug intake.
2. Male or female between 20 to 80 years old
3. Ability to provide written informed consent.

Exclusion Criteria:

1. Patients are still taking more than three anti-hypertensives at the screening visit
2. Pre-menopausal women
3. Known or suspected secondary hypertension
4. Mean sitting DBP<95mmHg and/or mean sitting SBP > 200mmHg at the end of placebo run-in phase
5. Hepatic and/or renal dysfunction
6. Known bilateral renal artery stenosis, patient with a solitary kidney, post renal transplant
7. Known NYHA functional class Chronic Heart Failure (CHF) III, IV
8. Unstable angina, myocardial infarction, cardiac surgery or stroke within the preceding six months
9. Post-Transluminal Coronary Angioplasty(PTCA) within the preceding three months
10. Sustained ventricular tachycardia, atria fibrillation, second or third degree AV block, VPC or APC (>10% of heart rate) or other clinically relevant cardiac arrhythmia as determined by the clinical investigator
11. Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of aortic or mitral valve.
12. Once documented evidence by ophthalmological examination of significant retinal haemorrhages/ exudates
13. Clinically significant sodium depletion as defined by serum sodium level less than 130 mmol/L
14. Clinically significant hyperkalemia as defined by serum potassium level >5.5 mmol/L
15. Non-insulin dependent DM poorly controlled whicih is defined as HbA1c>8% twice consecutively within 6 months and/or AC blood sugar>180 mg/dl.
16. Insulin Dependent Diabetes Mellitus
17. Chronic administration of oral anticoagulants and/or digoxin within the past 6 months.
18. Known drug or alcohol dependency
19. Administration of medication known to affect blood pressure, except medication allowed by the protocol
20. Angioedema with ACE inhibitors
21. Use of nitrates

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31
Dates: Start 2004-03; Primary Completion 2005-03 (Actual); Study Completion 2005-03

PRIMARY OUTCOMES:
Change from baseline in sitting diastolic blood pressure (DBP) at trough (24 hours post-dosing) at the last observation during the double-blind phase. | 8 weeks

SECONDARY OUTCOMES:
Change from baseline in sitting SBP, standing DBP, standing SBP, sitting and standing heart rate at trough as well as blood pressure control and blood pressure response as defined in study protocol at the last observation will be evaluated. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Taiwan Ltd.
Locations (1):
- Machay Memorial Hospital, Taipei, Taiwan